CLINICAL TRIAL: NCT05246813
Title: Metabolic Profiling of Hematopoietic Stem Cells in Clonal Hematopoiesis (CHIP): a Prospective Observational Study
Brief Title: Metabolic Profiling of Hematopoietic Stem Cells in Clonal Hematopoiesis (CHIP)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imelda Hospital, Bonheiden (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Michaël R Laurent, MD PhD, Principal Investigator, Imelda Hospital, Bonheiden
Other Study IDs: 20211214
Record Dates: First submitted 2022-02-10; First posted 2022-02-18 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Osteoporosis; Osteoarthritis, Hip; Hip Fractures; Clonal Hematopoiesis of Indeterminate Potential; Aging
MeSH Terms: conditions — Osteoporosis; Osteoarthritis, Hip; Hip Fractures | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood and bone marrow samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Osteoporotic hip fracture patients
  Interventions: Other: Blood and bone marrow cell collection
- Hip osteoarthritis patients
  Interventions: Other: Blood and bone marrow cell collection

INTERVENTIONS:
Other: Blood and bone marrow cell collection — Collection of blood and bone marrow

SUMMARY:
Bone marrow samples will be collected from patients undergoing hip arthroplasty surgery. Blood and bone marrow samples will be used for metabolic profiling and analysis of relevant CHIP mutations. Combined single-cell transcriptomics and mutation-specific single-cell genotyping (biotin-PCR using mutation-targeted primers followed by sequencing) will subsequently be performed. The gene expression profile of wildtype and mutant hematopoietic stem cells will be compared, performing both broad gene set enrichment analysis and targeted analysis of metabolic pathways.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older

Exclusion Criteria:

* known haematological condition (myelodysplasia, leukemia, cancer)
* inability to provide written informed consent

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing hip arthroplasty for hip osteoarthritis or osteoporotic hip fractures.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gene Set Enrichment Analysis (GSEA) Normalized Enrichment Score (NES) | One day

CONTACTS AND LOCATIONS:
Overall Officials: Nick Van Gastel, PhD, Principal Investigator — de Duve Institute
Locations (1):
- Imelda Hospital, Bonheiden, België, Belgium

IPD SHARING:
Plan to Share IPD: Undecided